CLINICAL TRIAL: NCT03588143
Title: Immediate Effects of Transcutaneous Electrical Nerve Stimulation and High Voltage Pulsed Stimulation on Subacromial Pain and Shoulder Movements
Brief Title: Immediate Effects of TENS and HVPS on Subacromial Pain and Shoulder Movements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Gürhan KARAKAYA (Other)
Collaborators: Muğla Sıtkı Koçman University (Other)
Responsible Party: Sponsor-Investigator, Mehmet Gürhan KARAKAYA, Principal investigator, Head of Neurological Rehabilitation Department, PT. PhD. Prof., Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 16/044
Record Dates: First submitted 2018-01-17; First posted 2018-07-17 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Shoulder Pain Chronic
Keywords: Subacromial pain; Joint range of motion; Electrotherapy; Physiotherapy; Impingement
MeSH Terms: interventions — Electric Stimulation; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Electrical stimulation with TENS (Active Comparator): TENS with 100 Hz frequency, 65 microseconds pulse duration, in continuous pattern
  Interventions: Device: Electrical stimulation
- Electrical stimulation with HVPS (Experimental): HVPS with twin spiked monophasic current at 100 pps frequency, in continuous pattern
  Interventions: Device: Electrical stimulation
- Placebo electrical stimulation (Placebo Comparator): same electrode placement with other interventions, using the same electrotherapy device, without activating the device except its time unit.
  Interventions: Device: Electrical stimulation

INTERVENTIONS:
Device: Electrical stimulation — Two kinds of electrical stimulation (TENS and HVPS) and placebo intervention
  Other Names: TENS; HVPS; Placebo

SUMMARY:
This study was performed to investigate the immediate effects of transcutaneous electrical nerve stimulation (TENS) and high voltage pulsed stimulation (HVPS) on resting pain and pain-free range of shoulder motion (pfROM) in patients with subacromial pain syndrome (SAPS).

DETAILED DESCRIPTION:
Transcutaneous electrical stimulation (TENS) and high voltage pulsed current/stimulation (HVPS) are both electrotherapeutic agents which can be used for pain relief in musculoskeletal conditions. Standard TENS devices usually deliver biphasic pulsed currents with a pulse duration between 50 μs and 1000 μs and pulse frequencies between 1 and 250 pps. HVPS devices are TENS-like devices which deliver direct current with twin monophasic spiked pulses of 10-500 V (500-ohm load) with a short pulse duration (microseconds). In both conventional TENS technique and HVPS for pain relief, the aim is to activate spinal gating mechanism by selectively stimulating large diameter Aβ fibers. Theoretically, high-frequency (~10-250 pps), low-intensity (nonpainful) currents are most efficient in selectively activating Aβ fibers, which is practically recognized by the user reporting 'strong but comfortable' nonpainful electrical paresthesia beneath the electrodes. There is no available evidence for the efficacy of TENS in patients with subacromial pain. Also, there has been little experimental work on the effects of HVPS on pain relief in the literature, as well as no known study for its efficacy in SAPS.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years-old
* Pain with active shoulder movements
* Subacromial pain for 2 weeks-2 months
* Positive Hawkins-Kennedy and painful arc tests, infraspinatus weakness; in addition to these, for patients with partial rotator cuff tear, a negative drop-arm test
* Neer stage 1-2

Exclusion Criteria:

* Radiologically confirmed malignity
* Acromial/acromioclavicular arthritis
* History of fracture or surgery in the affected shoulder-arm complex
* Clinically confirmed polyarthritis, rheumatoid arthritis, fibromyalgia, adhesive capsulitis or osteoarthritis of glenohumeral joint or subacromial region
* Cervical/thoracal spinal problem• Neurological problems which may affect upper extremity movements or pain perception (stroke, peripheral neuropathy, brachial plexus lesion, etc.)
* Neer stage 3 and indication for surgery
* Usage of analgesic medication
* Obesity (Body mass ≥30 kg/m2)
* Contraindications for TENS or HVPS
* Previous experience with electrophysical agents or physiotherapy
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change of pain-free shoulder range of motion | Change of pain-free shoulder range of motions from baseline at the end of 30 minutes of each intervention
  Pain-free ranges of active shoulder flexion, abduction, internal and external rotation were measured by a digital inclinometer (Baseline Digital Inclinometer, 2008 New York-USA), which was calibrated on a flat surface before each measurement. All evaluations were performed before and after each modality application. All of the measurements were performed by a physiotherapist blinded to the modalities applied (placebo/TENS/HVPS).

SECONDARY OUTCOMES:
Change of pain intensity | Change of pain intensity from baseline at the end of 30 minutes of each intervention
  The participants were asked to mark their resting pain intensity on a 0-10 cm visual analogue scale (VAS), where 0 cm indicated no pain and 10 cm indicated unbearable pain. The distance of the marked point from zero point was recorded as the intensity of pain. All evaluations were performed before and after each modality application. All of the measurements were performed by a physiotherapist blinded to the modalities applied (placebo/TENS/HVPS).

IPD SHARING:
Plan to Share IPD: Undecided